CLINICAL TRIAL: NCT03717441
Title: DNA Analysis of Discarded Media Drops From the Clinical IVF Cycles
Status: Recruiting | Type: Observational
Sponsor: Colorado Center for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Mandy Katz-Jaffe, PhD, Research Director, Colorado Center for Reproductive Medicine
Other Study IDs: 2018154
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Media drops form IVF cycle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: chromosome numeration of embryos — Use genomic technologies to analyze the discarded media drop for chromosome counting

SUMMARY:
Performing DNA analysis of discarded media drops from the clinical IVF cycles completed in our Center

DETAILED DESCRIPTION:
The purpose of this research study is to investigate for the presence of DNA in the surrounding media that is remaining after human clinical IVF cycles, to have a non-invasive way of obtaining markers of embryo chromosome numeration. Media recovered from the clinical IVF laboratory is typically discarded during an IVF cycle. Genomic technologies will be used to analyze the otherwise discarded media drop for chromosome counting.

ELIGIBILITY:
Inclusion Criteria:

* Any women undergoing an In Vitro Fertilization cycle (IVF) at the Colorado Center for Reproductive Medicine that is also having Comprehensive Chromosomal Screening (CCS) of embryos

Exclusion Criteria:

-

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruiting women undergoing In Vitro Fertilization with Comprehensive Chromosomal Screening of embryos
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
DNA Analysis of discarded media drops form the clinical IVF Cycles | 1 day
  Analyze media drop for presence of DNA to obtain embryo chromosome numeration

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Katz-Jaffe, PhD, Principal Investigator — Colorado Center for Reproductive Medicine
Locations (1):
- Colorado Center for Reproductive Medicine, Lone Tree, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided